CLINICAL TRIAL: NCT00032747
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind Trial to Evaluate the Effects of Vasopressin V2 Receptor Antagonist on Clinical Improvement in Patients With Severe Chronic Heart Failure
Brief Title: Safety Study of Vasopressin V2 Receptor Antagonist on Patients With Severe Chronic Heart Failure (AQUAVIT).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI4510; SR121463B
Record Dates: First submitted 2002-03-29; First posted 2002-04-01 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; Heart Disease
MeSH Terms: conditions — Heart Diseases

INTERVENTIONS:
Drug: Vasopressin V2 Receptor Antagonist

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group forced up-titration study. Randomization will be stratified according to the patient's baseline serum sodium concentration (137-144 and <137 mmol/L). The dose of study drug will be increased to the next level on Day 15, and the total duration of the double-blind treatment period is 120 days.

ELIGIBILITY:
* Men or women with chronic heart failure (NYHA Class IIIB and IV).
* Women must be post-menopausal or surgically sterilized; they cannot be pregnant or nursing.
* Age 21 to 80 years.
* Chronic heart failure of at least 3 months duration. For 2 months prior to screening, patients must have had symptoms at rest or on minimal exertion for more than 50% of the time. For 2 weeks prior to screening, patients must have had symptoms at rest or on minimal exertion for more than 90% of the time.
* Patients must be receiving a diuretic and an ACE inhibitor (or an angiotensin II receptor antagonist) for the treatment of heart failure.
* Patients may be receiving digoxin, a beta-blocker or spironolactone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2001-08; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Clinical status at day 120.

SECONDARY OUTCOMES:
NYHA functional class, left ventricular ejection fraction, global assessment,serum sodium concentration.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (9):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Emory University, Atlanta, Georgia
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Brian LGH Heart Institute, Lincoln, Nebraska
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - MUSC/Division Cardiology, Charleston, South Carolina
- Sanofi-aventis Administrative Office, Laval, Canada
- Sanofi-aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- See also: Related Info — http://www.centerwatch.com
- See also: Related Info — http://www.sanofi-aventis.com